CLINICAL TRIAL: NCT06460844
Title: Phase 1, Open-Label, Dose-Escalation Study to Evaluate Safety of a Single Intravitreal Injection of RTx-015 in Patients With Retinitis Pigmentosa or Choroideremia (ENVISION)
Brief Title: Study to Evaluate Safety of RTx-015 Injection in Retinitis Pigmentosa or Choroideremia Patients (ENVISION)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ray Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTx-015-CP-101
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Retinitis Pigmentosa; Choroideremia
MeSH Terms: conditions — Retinitis Pigmentosa; Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low Dose RTx-015 (Experimental): Single intravitreal injection of low dose RTx-015
  Interventions: Genetic: RTx-015
- Middle Dose RTx-015 (Experimental): Single intravitreal injection of middle dose RTx-015
  Interventions: Genetic: RTx-015
- High Dose RTx-015 (Experimental): Single intravitreal injection of high dose RTx-015
  Interventions: Genetic: RTx-015
- Higher Dose RTx-015 (Experimental): Single intravitreal injection of higher dose RTx-015
  Interventions: Genetic: RTx-015

INTERVENTIONS:
Genetic: RTx-015 — Intravitreal injection using gene therapy to deliver an optogenetic gene to the eye. Cells in the retina use this Optogenetic gene to make a protein that responds to light.

SUMMARY:
A Phase 1, open-label, non-randomized, dose-escalation study, where approximately 18 eligible patients with retinitis pigmentosa or choroideremia will be enrolled sequentially in up to 4 dose cohorts of RTx-015. Enrolled patients will receive a single, unilateral intravitreal injection of RTx-015 in the study eye at Visit 3 (Day 0) and be followed for a total of 5 years.

DETAILED DESCRIPTION:
This Phase 1, open-label, non-randomized, multicenter clinical trial is to evaluate the safety and preliminary efficacy of a single, uniocular intravitreal injection of an investigational optogenetic gene therapy, RTx-015, in patients with retinitis pigmentosa or choroideremia. Up to 4 dose cohorts are planned, and each cohort will consist initially of 3 patients. Eligible patients will be assigned to a dose cohort by sequential enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Informed consent obtained from the patient
* Clinical diagnosis of Retinitis Pigmentosa independent of causative mutation OR Clinical diagnosis of Choroideremia with known causative mutation
* Study eye and fellow eye Best Corrected Visual Acuity meeting study criteria
* Presence of retinal ganglion cells and/or retinal nerve fiber layer on Spectral Domain Optical Coherence Tomography testing at Screening confirmed by central image reading center
* Adequate organ function and general good health

Exclusion Criteria:

* Participation in a clinical study (ocular or non-ocular) with an investigational drug, agent, or therapy in the past six months
* Concurrent participation in another interventional clinical ocular study
* Prior receipt of any gene therapy (ocular or other), retinal implant, or ocular cell therapy
* Pre-existing eye conditions in either eye that would preclude the planned treatment or, in the opinion of the Investigator, are significant enough to interfere with the interpretation of study endpoints or procedural complications
* Known steroid responders if their intraocular pressure was not able to be managed effectively with topical pressure-lowering medications after prior use of steroid medications
* Complicating systemic diseases; complicating systemic diseases include those in which the disease itself, or the treatment for the disease, can alter ocular and/or Central Nervous System (CNS) function (e.g., radiation treatment of the orbit; leukemia with CNS/optic nerve involvement)
* Any immunological response dysfunction including, immuno-compromising diseases or use of immunosuppressive medications, among others
* Cataract or other ocular (including refractive) surgery, intraocular and/or peri-ocular injection in either eye within the prior four months (i.e., 120 days) prior to screening
* Prior vitrectomy or aphakia in the study eye
* Known sensitivity to any component of the study treatment or contraindication to medications planned for use in the peri-procedural period (e.g., povidone-iodine to prep for intravitreal injection)
* Known contraindication to prophylactic steroid regimen
* Current pregnancy or breastfeeding
* Any other condition that would not allow the patient to complete follow-up examinations during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 12 months
  The number of patients in each cohort with treatment-emergent adverse events categorized using MedDRA v24.0 or higher

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) at Month 6 and Month 12 | 6 and 12 Months
  Change from baseline to Month 6 and Month 12 after injection with RTx-015 in BCVA
Low Luminance Visual Acuity (LLVA) at Month 6 and Month 12 | 6 and 12 Months
  Change from baseline to Month 6 and Month 12 after injection with RTx-015 in LLVA
Multi luminance mobility at Month 6 and Month 12 | 6 and 12 Months
  Change from baseline to Month 6 and Month 12 after injection with RTx-015 in Visual Change from baseline to Month 6 and 12 in mobility performance at multiple luminance levels
Contrast Sensitivity at Month 6 and Month 12 | 6 and 12 Months
  Change from baseline to Month 6 and Month 12 after injection with RTx-015 in Contrast Sensitivity
Full-field static visual field testing at Month 6 and Month 12 | 6 and 12 Months
  Change from baseline to Month 6 and Month 12 after injection with RTx-015 in the total area in which objects can be seen
Low Vision Quality of Life at Month 6 and Month 12 | 6 and 12 Months
  Change from baseline in low vision quality of life at Month 6 and Month 12. An algorithm will be applied to assess a total score. Higher scores are a worsening of the condition.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - UCI Alpha Clinic, Orange, California
  - UPMC Vision Institute, Pittsburgh, Pennsylvania
  - Retina Consultants of Texas Research Centers, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: No